CLINICAL TRIAL: NCT04255550
Title: Hemodynamic Monitoring and Correlation Between Electrical Cardiometry and Esophageal Doppler in Patients Undergoing Major Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Collaborators: Theodor Bilharz Research Institute (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Other Study IDs: Hemodynamic monitoring
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Electrical Cardiometry VS Esophageal Doppler

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Esophageal doppler — It is a prospective observational clinical study to correlate hemodynamic monitoring between non-invasive Electrical Cardiometry and minimally invasive Esophageal Doppler during major abdominal surgery.
  Other Names: Electrical cardiometry

SUMMARY:
The aim of this study is to correlate hemodynamic monitoring between noninvasive Electrical Cardiometry and minimally invasive Esophageal Doppler in patients undergoing major abdominal surgery

DETAILED DESCRIPTION:
Cardiac output (CO) and Stroke Volume (SV) can be used as markers for global cardiovascular functions and can assess fluid responsiveness to ensure adequate tissue perfusion which is one of the essential concerns of anesthestists and intensivists The gold standard is the thermodilution procedure by pulmonary artery catheter (PAC), yet, cannot be considered as a routine owing to potential difficulty and virtual complications The development of safe, simple, minimally invasive or non-invasive techniques which estimate CO, SV and systemic vascular resistance (SVR) without invasive intravascular catheterization or dye injection is important for clinical decision-making and research in anesthesia and critical care medicine Echocardiography in comparison with other Doppler modalities is a potent diagnostic mean that has the superiority above the traditional PAC for both diagnostic precision and rapidity However, the use of echocardiography needs good training and relatively expensive. Another ultrasound based device is Esophageal Doppler(ED) which looks more suitable for prolonged hemodynamic monitoring. This technique is minimally invasive which calculates the blood flow velocity in descending aorta and can determine SV and CO with sound trustworthiness. Such technique needs less training than standard echocardiography or PAC Thoracic Electric Bioimpedance (TEB) is a noninvasive monitoring which correlates differences in thoracic electrical conductivity to thoracic aortic blood volume and flow. It is a simple method for detection of SV, CO, contractility, SVR, and thoracic fluid content (TFC) for continuous monitoring. The results of previous studies comparing impedance cardiography with thermo dilution and other methods like transoesophageal echocardiography (TEE) have been largely inconclusive which may referred to higher thorax fluid content and consequently higher conductivity after surgical procedure To overcome these problems, upgraded computer equipment and advanced algorithms are used in the newer model; electrical cardiometry (EC), that interprets the maximum changes in TEB and can calculate CO accurately in adults and neonates Although other study compared between two devices in patients undergoing major abdominal and pelvic surgeries , but the sample size was small rather than our study , also it included laparoscopic surgeries which affect hemodynamics (blood pressure , heart rate and other cardiac parameters ) in such points . In addition investigators used the old version of thoracic bio-impedance (NICOM) which is different from our device as we will us (ICON) , Like another study comparing between two devices used also the old version of thoracic bio-impedance and didn't specify the type of surgery at which the study was done . There are also other studies comparing the two devices one of them in paediatrics undergoing kasai operation and the second in patients during liver transplantation , these two studies contain two types of patients not included in the present study .

ELIGIBILITY:
Inclusion Criteria:

* Geriatric patients.
* American Society of Anesthesiologists (ASA) physical status II or III.
* Patients listed for elective major abdominal surgery such as (e.g. cancer stomach, colon, bladder, or pancreas).

Exclusion Criteria:

* Age <50 years.
* Patients with hemodynamic instability and on inotropes which means ( perfusion failure, represented by clinical features of circulatory shock and advanced heart failure , It may also be defined as 1 or more out-of-range vital sign measurements, such as low blood pressure).
* Coagulopathies (platelet < 100×109/L, PT > 16 s and INR > 1.2).
* History of esophageal pathology.
* Patient needed massive blood transfusion intraoperatively which means replacement of >1 blood volume in 24 hours or >50% of blood volume in 4 hours (adult blood volume is approximately 70 mL/kg).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Demographic data, hemodynamic parameters as heart rate (HR), and mean arterial blood pressure (MAP), and urine output will be registered.
  Cardiac data derived from EC and ED including: CO ,cardiac index( CI), SV, stroke volume index( SVI),systemic vasculare resistance (SVR), and oxygen delivery index (DO2I) will be also recorded.
  Cardiac data will be recorded at the following time:
  1. T1 baseline: prior to skin incision.
  2. T2: one hour after induction.
  3. T3: half an hour after organ resection.
  4. T4: at the end of surgical procedure. During arrhythmias or hemodynamic instability, measurements will not be recorded.
  After the end of surgery, muscle relaxation will be reversed with 0.05 mg/kg neostigmine and 0.02 mg/kg atropine. Postoperative pain relief will be achieved by intravenous administration of 1mg/kg mepridine and 1gm acetaminophen every 12 hours.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Cardiac Output measurement | 24 hours Postoperative
  Correlation between two devices regarding Cardiac Output measurement

SECONDARY OUTCOMES:
Cardiac Index | Up to 24 hours
  Assessment of other hemodynamic parameter Cardiac Index
Stroke Volume | Up to 24 hours
  Assessment of other hemodynamic parameter Stroke Volume
Stroke Volume Index | Up to 24 hours
  Assessment of other hemodynamic parameter Stroke Volume Index
Syetemic Vascular Resestance | Up to 24 hours
  Assessment of other hemodynamic parameter Syetemic Vascular Resestance

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Kaddah, M.D, Principal Investigator — Cairo University; Abla Elhadedy, M.D, Principal Investigator — Theodor Bilharz Institute; Shady Rady Abdalla, M.D, Principal Investigator — Cairo University; Ahmed salah abdelazeem elsayed, M.Sc., Principal Investigator — Theodor Bilharz Institute; Ahmed Abdalla Mohamed, M.D, Study Chair — Cairo University; Hanan Khafagy, M.D, Study Director — Theodor Bilharz Institute; Reham Saeed, M.D, Study Director — Theodor Bilharz Institute; Haitham Abouzeid, M.D, Study Director — Theodor Bilharz Institute; Ahmed Essam, M.D, Study Director — Theodor Bilharz Institute
Locations (1):
- Tarek Kaddah, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till Publication